CLINICAL TRIAL: NCT03563326
Title: Clinical Trial of Intraperitoneal CAR-T Cells Infusion for the Treatment of Advanced Gastric Cancer With Peritoneal Metastasis
Brief Title: Intraperitoneal Infusion of EpCAM CAR-T Cell in Advanced Gastric Cancer With Peritoneal Metastasis (WCH-GC-CART)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jian-Kun Hu (Other)
Responsible Party: Sponsor-Investigator, Jian-Kun Hu, Vice director of Gastrointestinal Surgery department, West China Hospital; Director of Institute of Gastric Cancer, State Key Laboratory of Biotherapy, West China Hospital, West China Hospital
Organization: West China Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WCH-GC-CART
Record Dates: First submitted 2018-05-05; First posted 2018-06-20 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2018-09

CONDITIONS: Neoplasm, Stomach; Metastases, Neoplasm; Neoplasm Seeding
Keywords: Epithelial Cell Adhesion Molecule; Chimeric Antigen Receptor-modified T cell; Gastric carcinoma; Peritoneal metastasis
MeSH Terms: conditions — Stomach Neoplasms; Neoplasm Metastasis; Neoplasm Seeding; Colorectal Cancer, Hereditary Nonpolyposis, Type 8 | interventions — Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CAR-T cell and chemotherapy (Experimental): Biological: CAR-T cells targeting EpCAM Chemotherapy: determined by medical Oncologist
  Interventions: Biological: CAR-T cells targeting EpCAM; Biological: Chemotherapy
- chemotherapy (Active Comparator): Chemotherapy: determined by medical Oncologist
  Interventions: Biological: Chemotherapy

INTERVENTIONS:
Biological: CAR-T cells targeting EpCAM — Biological: CAR-T cells targeting EpCAM
  Arms: CAR-T cell and chemotherapy
Biological: Chemotherapy — Chemotherapy: determined by medical Oncologist

SUMMARY:
To investigate the safety and efficacy of intraperitoneal infusion of EpCAM CAR-T cell in advanced gastric cancer with peritoneal metastasis by a prospective nonrandomized controlled trial.

DETAILED DESCRIPTION:
Chimeric antigen receptor modified T (CAR-T) cells have the capability in targeting and recognizing tumor antigen, and can specifically recognize, bind and kill tumor cells with positive antigen. Through local drug delivery, CAR-T cells have successfully achieved remarkable effect to treat solid tumors. Gastric cancer is one of the most frequent malignant tumors with high mortality, especially in China. Peritoneal metastasis is one of the common routes of metastasis. Once peritoneal metastasis occurred, patients should be categorized as clinical pathological stage IV with extremely poor prognosis, and the effect of routine treatments would be unsatisfactory. Epithelial cell adhesion molecule (EpCAM) is highly expressed in gastric cancer cells and closely associated with the poor prognosis of patients. In our previous pre-clinical research researches, the investigators have obtained CAR-T cells targeting EpCAM (EpCAM CAR-T), and finished the preparations of cells which could be used in clinical practice. Based on our previous works, the investigators aim to investigate the safety and efficacy of peritoneal infusion of EpCAM CAR-T cell in advanced gastric cancer with peritoneal metastasis by a prospective nonrandomized controlled trial. The results of this clinical trial are expected to provide the new treatment strategy for gastric cancer patients with peritoneal metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with EpCAM positive gastric cancer who have peritoneal metastasis at first visit; Patients with highly suspected or previous proven peritoneal metastasis by biopsy, CT, digital rectal examination, etc. who failed to the routine therapies like chemotherapy;
2. Age between 18 and 75;
3. Estimated survival time is longer than 3 months;
4. Eastern Cooperative Oncology Group (ECOG）scores 0-2;
5. Hemoglobin≥90g/L, ANC≥1.5×109/L, PLT≥80×109/L;
6. Negative pregnancy test for child-bearing period; both male and female patients should agree to apply effective contraceptive methods in the period of treatment and one year after treatment;
7. Both patients and families totally understand the objectives and risks of the treatments and sign the informed consent.

Exclusion Criteria:

1. Comorbidity with other diseases treated by immunosuppressive drugs or steroids therapy systematically;
2. Uncontrolled active infection;
3. HIV positive;
4. Active hepatic B or C virus infection, active tuberculosis;
5. Pregnant or lactation female;
6. Disagree to apply effective contraceptive methods in the period of treatment and one year after treatment;
7. Positive cytology examination alone.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-08-30 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
EpCAM CAR-T cells treatment related adverse events | 4 weeks
  Adverse events after receiving EpCAM CAR-T cells treatment, according to NCI-CTCAE v4.0.

SECONDARY OUTCOMES:
Overall survival outcome | 2 years
  2-year overall survival rate
Metabolism kinetics of CAR-T cells | 2 years
  The level of CAR-T cells will be tested regularly by Real-time Quantitative Polymerase Chain Reaction Detecting System(qPCR) or Flow cytometry.
Progress free survival outcome | 2 years
  2-year progress free survival

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Kun Hu, M.D. Ph.D., Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided
pending